CLINICAL TRIAL: NCT05518799
Title: Phenotyping Study of CYP3A4 Activity in Patients With Prostate Cancer Versus Male Patients With Other Types of Solid Tumours With Midazolam
Brief Title: CYP3A4 Activity in Patients With Prostate Cancer Versus Male Patients With Other Solid Tumours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: N20CYM
Record Dates: First submitted 2022-07-15; First posted 2022-08-29 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer; Solid Tumor, Adult
Keywords: midazolam; CYP3A4; pharmacokinetics; phenotyping
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with prostate cancer (Other)
  Interventions: Drug: Midazolam
- Male patients with other types of solid tumours (Other)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — Patients will receive 2 mg midazolam orally on day 1 of the study and 1 mg midazolam intravenously on day 2 of the study.

SUMMARY:
The hepatic enzyme, cytochrome P450 3A4 (CYP3A4) is important for the metabolism of many drugs including taxanes. Previous reported studies reported a decreases in docetaxel exposure in prostate cancer patients compared to patients with other solid tumours. The difference was 1.8-fold for intravenous administration and 2.8-fold for oral administration.

The underlying mechanism for these observations remains to be elucidated. The lower docetaxel exposure with IV and oral docetaxel treatment might be related to a higher CYP3A4 activity in prostate cancer patients. Therefore, it is important to directly compare the CYP3A4 activity with a phenotyping test in prostate cancer patients and patients with other types of solid tumours.

This is an in vivo phenotyping studying using midazolam as a probe for CYP3A4 activity in patients with prostate cancer and patients with other solid tumours. The primary objective is the comparison of CYP3A4 activity in prostate cancer patients versus male patients with other types of solid tumours by use of an oral midazolam phenotyping test. Secondary objectives are: (1) measurement of plasma concentrations of midazolam and it's two primary metabolites (1'-hydroxy midazolam and 4'-hydroxy midazolam), (2) determination of the metabolite pharmacokinetics of midazolam. (3) retrospective assessment of single nucleotide polymorphisms of CYP3A4. The exploratory objective is to differentiate between gastro-intestinal and hepatic CYP3A4 activity with oral and intravenous administration of midazolam.

DETAILED DESCRIPTION:
The metabolizing enzyme cytochrome P450 (CYP) 3A4 is an important factor in the pharmacokinetics (PK) of many (anticancer) drugs, including taxanes [1]. Recently, it has been reported that the PK of intravenous docetaxel are different in patients with castration resistant prostate cancer, as compared to patients with other types of solid tumours [2]. Different phase I studies with the oral docetaxel formulation ModraDoc006 in combination with ritonavir (denoted as ModraDoc006/r), were conducted in our institute in patients with hormone-sensitive prostate cancer (HSPC), metastatic castration-resistant prostate cancer (mCRPC) and other types of solid tumours [3-5]. The exposure to docetaxel and ritonavir after administration of the same dose and schedule of ModraDoc006/r was substantial lower in prostate cancer patients as compared to the patients with other types of solid tumours. In contrast to the 1.8-fold difference reported with IV docetaxel, the difference in the area under the plasma concentration versus time curve (AUC) was 2.8-fold with oral ModraDoc006/r treatment [2-5]. The PK-curves of docetaxel and ritonavir are shown in figure 1A and 1B.

The underlying mechanism for these observations remains to be elucidated. The lower docetaxel exposure with IV and oral docetaxel treatment and the lower ritonavir exposure with ModraDoc006/r treatment might be related to a higher CYP3A4 activity in prostate cancer patients. Therefore, it is important to directly compare the CYP3A4 activity with a phenotyping test in prostate cancer patients and patients with other types of solid tumours.

As a potential cause for this, CYP3A4 activity might be altered by medical castration. Franke et al. showed that the clearance of docetaxel was higher in castrated versus non-castrated prostate cancer patients. However, comparison of the CYP3A4 activity in the castrated versus the prostate cancer patients with normal levels of testosterone showed no significant differences [6]. However, this was done in 6 CRPC patients, of which one patient had an extremely low CYP3A4 activity. The intravenous erythomycin breath test that was used in this study only reflects the hepatic CYP3A4 activity and not the gastro-intestinal CYP3A4 activity. The latter is important in treatment with oral docetaxel (ModraDoc006) in combination with ritonavir. Furthermore, erythomycin is also a substrate for P-glycoprotein (P-gp), indicating that the erythomycin breath test might reflect P-gp activity as well as CYP3A4 activity [7,8]. Therefore, it is necessary to evaluate prostate cancer patients with a phenotyping test that includes both the hepatic and gastro-intestinal CYP3A4-activity.

Midazolam is one of the most frequently used test compounds used for evaluation of CYP3A4 activity [9-11]. Midazolam has several advantages over other CYP3A4 probes such as erythromycin, dapsone, quinine, and nifedipine [11]. First, midazolam is selectively metabolized by CYP3A4 [9,10]. Furthermore, midazolam clearance after both oral and intravenous administration is a widely accepted and validated metric of CYP3A4 activity [9-11]. Continuing, midazolam AUC and metabolite clearance to its major metabolite 1-hydroxy midazolam correlate well with hepatic CYP3A content [11-13]. Also, midazolam PK are highly sensitive to changes in CYP3A4 activity [9-11]. Therefore, oral midazolam will be used in this study to further evaluate the CYP3A4 activity in prostate cancer patients in comparison to patients with other types of solid tumours. To further differentiate between gastro-intestinal and hepatic CYP3A4 activity, evaluation with both oral and intravenous midazolam is included in this study.

1. Mathijssen RHJ, van Schaik RHN. Genotyping and phenotyping cytochrome P450: perspectives for cancer treatment. Eur J Cancer 2006; 42(2):141-8
2. De Vries Schultink AHM, Crombag MBS, van Werkhoven E, et al. Neutropenia and docetaxel exposure in metastatic castration-resistant prostate cancer patients: A meta-analysis and evaluation of a clinical cohort. Cancer Med 2019; 8(4): 1406-15.
3. De Weger VA, Stuurman FE, Hendrikx J, et al. A dose-escalation study of bi-daily once weekly oral docetaxel either as ModraDoc001 or ModraDoc006 combined with ritonavir. Eur J Cancer 2017; 86: 217-25.
4. Vermunt MAC, Janssen JM, Vrijenhoek GL, Van der Poel HG, Thijssen B, Beijnen JH et al. Addition of an oral docetaxel treatment (ModraDoc006/r) to androgen deprivation therapy (ADT) and intensity-modulated radiation therapy (IMRT) in patients with high risk N+M0 prostate cancer. Ann Oncol 2019; 30(suppl_5): v325-v355
5. Vermunt M, Robbrecht D, Devriese L, Janssen J, Keessen M, Eskens F et al. ModraDoc006, an oral docetaxel formulation in combination with ritonavir (ModraDoc006/r), in metastasized castration-resistant prostate cancer (mCRPC): A multicenter phase I study. J Clin Oncol. 2020; 38(suppl 6;abstr 79)
6. Franke RM, Carducci MA, Rudek MA, Baker SD, Sparreboom A. Castration-dependent pharmacokinetics of docetaxel in patients with prostate cancer. J Clin Oncol. 2010 Oct;28(30):4562-7
7. Lan LB, Dalton JT, Schuetz EG. Mdr1 limits CYP3A metabolism in vivo. Mol Pharmacol 2000;58:863-9
8. Chiou WL, Chung SM, Wu TC. Potential role of P-glycoprotein in affecting hepatic metabolism of drugs. Pharm Res 2000;17:903-5.
9. Streetman DS, Bertino JS, Nafziger AN. Phenotyping of drug-metabolizing enzymes in adults: a review of in-vivo cytochrome P450 phenotyping probes. Pharmacogenetics 2000; 10(3):187-216
10. Hohmann N, Haefeli WE, Mikus G. CYP3A activity: towards dose adaptation to the individual. Expert Opin Drug Metab Toxicol 2016; 12(5):479-97
11. Fuhr U, Jetter A, Kirchheiner J. Appropriate phenotyping procedures for drug metabolizing enzymes and transporters in humans and their simultaneous use in the "cocktail" approach. Clin Pharmacol Ther 2007; 81(2): 270-83
12. Thummel KE, Shen DD, Podoll TD, Kunze KL, Trager WF, Hartwell PS et al. Use of midazolam as a human cytochrome P450 3A probe: I. In vitro-in vivo correlations in liver transplant patients. J Pharmacol Exp Ther 1994; 271(1):549-56
13. Thummel KE, Shen DD, Podoll TD, Kunze KL, Trager WF, Bacchi CE et al. Use of midazolam as a human cytochrome P450 3A probe: II. Characterization of inter- and intraindividual hepatic CYP3A variability after liver transplantation. J Pharmacol Exp Ther 1994; 271(1):557-66

ELIGIBILITY:
Inclusion Criteria:

1. Male patients receiving anticancer treatment or supportive care within our institute

   * Group 1: histological or cytological proof of prostate cancer, for which the treatment leads to castrate levels of testosterone. Both metastatic as non-metastatic patients can be included. Both hormone-sensitive as castration-resistant patients can be included. Castrate levels of testosterone are defined as ≤ 50 ng/dL (or ≤ 0.50 ng/mL or 1.73 nmol/L)
   * Group 2: men with histological or cytological proof of cancer. Both metastatic as non-metastatic patients can be included.
2. Considered fit for midazolam treatment as assessed by the treating physician.
3. Age ≥ 18 years.
4. Able and willing to give written informed consent.
5. Able and willing to undergo blood sampling for PK and pharmacogenetic analysis.
6. Able and willing to comply with study restrictions and to remain at the study center for the required duration. The obligated duration is up to 8 hours after oral administration of midazolam on day 1. Day 2 has a duration of 8 hours after the intravenous administration of midazolam.
7. Adequate organ system function as defined as:

   * Absolute neutrophil count equal or greater than 1.5x 10^9 /L
   * Hemoglobin equal or greater to 6.0 mmol/L
   * Platelets greater or equal to 100 x 10^9 /L
   * Total bilrubin equal or smaller than 1.5 x ULN
   * AST and ALT equal or smaller than 2.5 x ULN
   * Serum creatinine clearance equal or smaller of 1.5 x ULN or eGRF greater or equal to 40 mL/min determined by de MDRD-4.

Exclusion Criteria:

1. Concomitant use of medication, herbs or food which could influence the pharmacokinetics of midazolam within 14 days or five half-lives of the drug (whichever is shorter) before start of the study, consisting of (but not limited to) CYP3A4-inhibitors/inducers. In particularly, bicalutamide and dexamethasone are not allowed within 14 days before start of the study. The use of enzalutamide is prohibited within 30 days before start of the study. The use of prednisolone is allowed before and during the study at a maximum daily dose of 10 mg.
2. Current smokers or patients who stopped smoking within 7 days before study allocation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
CYP3A4 | One study day
  Midazolam clearance is a generally accepted biomarker for CYP3A4 actiivty

SECONDARY OUTCOMES:
Measurement of plasma concentrations of midazolam, 1'-hydroxy midazolam and 4'-hydroxy midazolam | through study completion, an average of 1 year
  Plasma concentrations will be determined with LC-MS/MS. The unit will be microgram/L.
Pharmacokinetics of midazolam, 1'-hydroxy midazolam, and 4'-hydroxymidazolam | through study completion, an average of 1 year
  Non-lineair mixed effects modelling (NONMEM) will be performed to determine the pharmacokinetic profile
Single nucleotide polymorphisms in the genes encoding for CYP3A4 | through study completion, an average of 1 year
  polymerase chain reaction to identify single nucleotide polymorphisms in the genes encoding for CYP3A4

OTHER OUTCOMES:
Differentiation between gastro-intestinal and hepatic CYP3A4 activity with oral and intravenous administration of midazolam. | through study completion, an average of 1 year
  Non-linear mixed effects modelling (NONMEM) will be performed to determine the contribution of hepatic CYP3A4 content and gastro-intestinal CYP3A4 concent on midazolam clearance.

CONTACTS AND LOCATIONS:
Overall Officials: F Opdam, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek/The Netherland Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No